CLINICAL TRIAL: NCT07007871
Title: Evaluating the Impact of a Tutoring and Counseling Program for Low Income Secondary School Students With Mental Challenges in Hong Kong During COVID-19: A Randomized Control Trial
Brief Title: Mindmatters: Tutoring and Counseling Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EdUHK Mindmatters
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Issues
Keywords: Adolescents; counselling; mental health; tutoring; pandemic
MeSH Terms: conditions — Psychological Well-Being | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: A randomized waitlist-controlled design will be used to examine the effectiveness of the tutoring and counseling service program. Eligible secondary school students will be allocated to the experimental group and waitlist control group, alongside trained university student tutors with education or psychology background. All assessments will be conducted individually for each student by independent assessors who are blinded to the treatment conditions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Students allocated to the experimental group begin receiving the tutoring and counseling program.
  Interventions: Other: Tutoring and Counselling (1)
- Waitlist Control Group (Other): Students assigned to the waitlist control group receive the program after the experimental group completes it.
  Interventions: Other: Tutoring and Counselling (2)

INTERVENTIONS:
Other: Tutoring and Counselling (1) — During the intervention, students participate in a structured program designed to support those with confirmed or suspected mental illness. The program includes two weekly group tutorial sessions lasting 1.5 hours each, organized in small groups of 4-5 students to foster interaction and peer support. Students also receive two individual counseling sessions per month, each lasting one hour. Tutor-group assignments are based on tutor availability and location for logistical efficiency.
  Arms: Experimental Group
Other: Tutoring and Counselling (2) — Students assigned to the waitlist control group receive the program after the experimental group completes it. Students participate in a structured program designed to support those with confirmed or suspected mental illness. The program includes two weekly group tutorial sessions lasting 1.5 hours each, organized in small groups of 4-5 students to foster interaction and peer support. Students also receive two individual counseling sessions per month, each lasting one hour. Tutor-group assignments are based on tutor availability and location for logistical efficiency.
  Arms: Waitlist Control Group

SUMMARY:
The tutoring and counseling program for adolescents from low socioeconomic backgrounds facing mental health challenges during the COVID-19 pandemic will be assessed using a randomized controlled trial. The study will recruit secondary students with confirmed or suspected mental illnesses and trained university student tutors with backgrounds in education or psychology. The program provides both online and in-person support. Various measures, including surveys on depression, anxiety, stress, academic performance, executive function, emotional and behavioral issues, and tutor efficacy, will be used. Qualitative feedback will be gathered through open-ended questions. It is hoped that the findings will contribute valuable insights into effective support strategies for this vulnerable population.

DETAILED DESCRIPTION:
The COVID-19 pandemic significantly affected the academic performance and mental well-being of adolescents, especially those facing both low socioeconomic status (SES) and mental health challenges. Research shows that disparities in educational access experienced from low SES families were exacerbated four times by the shift to remote learning during the pandemic. This lack of access to essential technology and conducive learning environments, further impeding their academic progress and mental well-being. Additionally, the pandemic intensified the mental health struggles of this group of vulnerable adolescents, leading to increased feelings of isolation, uncertainty, and anxiety. Such profound impact of the pandemic underscores the critical need for comprehensive support in both academic performance and mental well-being. It is imperative to adopt a holistic approach that addresses both dimensions.

This study evaluates the effectiveness of an innovative tutoring and counseling program. This program involves university students who have undergone 39 hours of training, serving as tutors to provide online and face-to-face support to low SES adolescents with mental health challenges. To equip the university students for their roles, a web-based online training platform was developed by the first author. This platform includes 14 courses, each comprising a) teaching video clips by the course lecturer, b) relevant reading materials in Chinese and English, and c) 1-2 online quizzes. The content of these modules covers effective pedagogies, counseling and psychotherapy, and mental health knowledge, ensuring that the tutors are well-prepared to address the diverse needs of the adolescents they support. This paper begins by discussing the exacerbated academic disparities and mental health challenges encountered by this targeted group amid the COVID-19 pandemic. Subsequently, it investigates the unique challenges faced by this group of adolescents in Hong Kong (HK) and the need for a comprehensive intervention program tailored to their specific needs.

During the pandemic, the extended closure of schools and strict social distancing measures worsened the psychosocial well-being of adolescents. This impact extended to various social aspects, including compromised learning opportunities, diminished social relationships and connectedness, and heightened concerns about the pandemic, coupled with a sense of financial insecurity. In particular, the pandemic has disproportionately affected adolescents coming from low SES backgrounds. These challenges, arising from a combination of economic disparities and disruptions in educational paradigms, have significantly compromised both academic performance and overall well-being within this demographic cohort. Early in the pandemic, Kuhfeld et al. estimated that students from marginalized backgrounds would experience more pronounced academic setbacks, diverting them further from their educational objectives. Previous study substantiates this claim, revealing that disruptions induced by the pandemic in the education system led to substantial learning regression, particularly affecting students from low SES backgrounds.

In fact, adolescents from low SES backgrounds undeniably encounter significant impediments in accessing educational resources and opportunities, encompassing essential technology, stable internet connections, or conducive learning environments. A recent study by Agostinelli et al. scrutinized the impact of school closures on student learning, revealing that students from lower-income households experienced more profound learning losses as compared to their more affluent peers, signifying an exacerbation of educational disparities post-pandemic. A study in Australia revealed that during the pandemic, the achievement gap widens threefold in remote schooling compared to traditional classrooms. Even when remote learning is effective, students facing disadvantages are estimated to progress at approximately 50 percent compared to their affluent peers.

Moreover, the regression in learning has further intensified stress within this demographic group, amplifying their sense of inadequacy and frustration. A recent investigation in HK suggested that adolescents with lower SES face heightened vulnerability to psychosocial distress during the pandemic due to increased difficulties in learning and a sense of isolation. Dawson and Golijiani-Moghaddam proposed that students from low SES bear a disproportionate burden, with an elevated likelihood of experiencing challenges such as food insecurity and housing instability during the pandemic, further complicating their mental health issues. The intricate interplay of the pandemic's effects on academic disparities and mental well-being among adolescents with low SES underscores the necessity for targeted interventions and the establishment of comprehensive support frameworks.

Undoubtedly, for students already facing suspected or confirmed mental health issues, the pandemic significantly intensified their struggles. Research by Hafstad et al. reported a significant increase in symptoms of depression and anxiety among students, particularly those already dealing with pre-existing mental health issues. Many studies confirmed that individuals with pre-existing mental health conditions might be particularly susceptible to heightened emotional stress triggered by the pandemic, potentially leading to relapses or a deterioration of their mental well-being. Furthermore, mental health services available to patients were restricted due to the demands of the pandemic. Some individuals experienced extended follow-up periods to minimize virus exposure, while community centers were temporarily closed in adherence to social distancing policies. A World Health Organization survey across 130 countries revealed that, despite an increasing demand, critical mental health services were disrupted or halted in 93% of countries globally. As a result, individuals who required assistance mostly received inadequate support during the COVID-19 outbreak, despite the clear and pressing needs.

In addition to the insufficient well-being support, the deterioration of mental well-being amid the COVID-19 pandemic has manifested in diverse ways that further affect academic performance in a group of low SES adolescents. The deterioration of mental well-being not only intensifies academic regression within this demographic group but also casts a shadow on cognitive functions, especially executive functions. Research indicates that students struggling with declining mental health often face challenges in concentration and inhibitory control, leading to difficulties in suppressing attention to irrelevant input. Elevated stress and anxiety levels can further impede working memory, contributing to struggles in managing workloads. Moreover, studies suggest that the presence of depressive moods and disrupted sleep hinder effective problem-solving skills and cognitive flexibility. More importantly, all these cognitive deficits collectively contribute to further impediments in academic performance and mental health.

Additionally, social isolation and a lack of social support contribute to a sense of disconnection, impacting attendance, active participation, and overall engagement in academic activities for this group of already vulnerable adolescents. This intricate interplay among insufficient mental health support, cognitive setbacks, and academic regression underscores the critical need to comprehensively address the well-being of these young individuals. It emphasizes the necessity for supportive measures that encompass both academic and well-being aspects to foster a conducive environment for their growth and development.

Until February 2022, HK demonstrated effective containment of the pandemic, albeit under the imposition of stringent social distancing measures. Diverging from the relatively shorter school closures in Western counterparts, secondary school students in HK endured an extended period of more than two years marked by intermittent episodes of remote learning. This protracted duration deprived them of sustained educational, social, and emotional support tailored to their specific needs. Moreover, HK's unique socio-environmental features, characterized by a low average living area per capita (13.8 square meters per person) disproportionately affected adolescents from low-income families.

In fact, empirical investigations highlight the positive correlation between residing in densely populated environments with restricted access to outdoor spaces and heightened levels of depression during the pandemic. The heightened risk of community-acquired infections in densely populated regions further contributed to pandemic-related stress. Concurrently, elevated stress levels experienced by parents also exerted a deleterious influence on the adjustment of their teenage children. Epidemiological data from 2022 underscored the prevalence of mild to extremely severe depression (39.6%), anxiety (37.5%), and stress (48.8%) among adolescents in HK, particularly poignant for those contending with limited resources and mental health complexities. The distinctive challenges faced by adolescents in this densely populated locale amid the COVID-19 pandemic warrant meticulous consideration and targeted interventions.

It is crucial to recognize that undergraduate students also faced significant challenges during the pandemic. Many of them had to adapt to online learning environments and cope with the lack of exposure to practical experiences. Research by Nicholson et al. documented that university students experienced increased stress and reduced motivation due to the abrupt transition to online classes. The absence of in-person interactions with teachers and peers also posed challenges for their academic and social development. Moreover, university students were affected by the limited access to extracurricular activities, internships, and hands-on learning opportunities, which are integral to their holistic development. The disruption of these essential aspects of their educational journey underlines the importance of providing targeted support to help them effectively acquire skills and gain valuable experiences in order to navigate these challenges.

The pandemic has unleashed a profound and multifaceted impact on students confronting mental health challenges within low SES background. Academic disparities have been exacerbated, learning loss has become pervasive, and mental health struggles have intensified. As the pandemic evolves, the urgency to address these challenges becomes increasingly apparent. In response to these formidable challenges, the current study evaluates the effectiveness of a pioneering tutoring and counseling program, named "Mind and Study Matter". This initiative aims to train university students from education-related or psychology-related disciplines as tutors. These tutors provide both online and face-to-face support to low SES students with suspected mental difficulties in secondary schools. Extensive research underscores the high effectiveness of peer tutoring in enhancing academic outcomes. This innovative approach not only recognizes the distinct ability of university students to connect with their peers but also acknowledges the heightened demand for support in the post-pandemic landscape.

Indeed, the exposure and training offered through tutoring programs have been shown to significantly enhance tutors' self-efficacy in inclusive education. Research by Johnson found that undergraduate students engaged in tutoring programs demonstrated increased confidence in their ability to support diverse learners. Evidence from Strawbridge et al. further supports this, emphasizing that hands-on experience in tutoring sessions, coupled with targeted training modules, positively influenced tutors' beliefs in their capacity to cater to the educational needs of a diverse student population.

Moreover, tutoring program exposure has been associated with increased empathy and understanding among tutors regarding the challenges faced by marginalized students. This exposure, combined with knowledge in inclusive practices, is confirmed to improve the ability to create supportive and inclusive learning environment.

In addition, tutoring programs have proven to be indispensable, especially in the context of the pandemic, in addressing the academic disparities and learning setbacks faced by students from low SES backgrounds. Abundant research attests to the transformative impact of tutoring, effectively bridging educational gaps and alleviating academic setbacks. The personalized guidance offered by tutors is instrumental in restoring confidence and academic progress among students with low SES, helping them bridge the educational gap with their peers. Furthermore, the integration of mental health support within tutoring programs aligns seamlessly with the growing recognition of the interconnectedness of academic and mental health challenges. Tutors play a pivotal role in providing emotional guidance and fostering a supportive environment, effectively addressing the amplified stress and anxiety experienced by students during the pandemic. Moreover, through thorough training and supervised guidance, the incorporation of university students as tutors in this initiative constitutes a valuable asset for providing academic support and mentorship.

ELIGIBILITY:
Inclusion Criteria:

* aged between 12 and 18 years
* studying at secondary schools in HK
* low socioeconomic status
* confirmed or suspected mental illness

Exclusion Criteria:

* diagnosed with neurological needs
* received tutoring and counselling

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Depression, anxiety, and stress | One week before the intervention
  The Depression, Anxiety and Stress Scale (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains seven items, divided into subscales with similar content. Students are asked to rate on a 4-point Likert scale from 0 (never) to 3 (almost always).
Depression, anxiety, and stress | One week after the intervention
  The Depression, Anxiety and Stress Scale (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains seven items, divided into subscales with similar content. Students are asked to rate on a 4-point Likert scale from 0 (never) to 3 (almost always).
Executive function | One week before the intervention
  The Behavior Rating Inventory of Executive Function (BRIEF) is designed to assess executive function in the home environment. A short version of the BRIEF consists of nine items, with the following three scales obtained: Working memory, inhibition, and cognitive flexibility. Parents are asked to rate their child's behavior on a 3-point Likert scale ranging from 1 (never) to 3 (often).
Executive function | One week after the intervention
  The Behavior Rating Inventory of Executive Function (BRIEF) is designed to assess executive function in the home environment. A short version of the BRIEF consists of nine items, with the following three scales obtained: Working memory, inhibition, and cognitive flexibility. Parents are asked to rate their child's behavior on a 3-point Likert scale ranging from 1 (never) to 3 (often).
Conduct problem and emotional symptoms | One week before the intervention
  The emotional symptoms and conduct problems subscales of the Strengths and Difficulties Questionnaire (SDQ) are administered to parents to assess the child's behavior over the last six months. Each subscale consists of five items using a 3-point Likert scale: 0 (not true), 1 (somewhat true), and 2 (certainly true). Higher scores reflect more severe difficulties.
Conduct problem and emotional symptoms | One week after the intervention
  The emotional symptoms and conduct problems subscales of the Strengths and Difficulties Questionnaire (SDQ) are administered to parents to assess the child's behavior over the last six months. Each subscale consists of five items using a 3-point Likert scale: 0 (not true), 1 (somewhat true), and 2 (certainly true). Higher scores reflect more severe difficulties.
Teacher-reported academic achievement | One week before the intervention
  Students' academic achievement in Chinese, English, and Mathematics is rated by teachers using a 5-point scale. The scale ranged from 1 (bottom 20% of the performance) to 5 (top 20% of performance).
Teacher-reported academic achievement | One week after the intervention
  Students' academic achievement in Chinese, English, and Mathematics is rated by teachers using a 5-point scale. The scale ranged from 1 (bottom 20% of the performance) to 5 (top 20% of performance).
Parental stress | One week before the intervention
  The Parental Stress Scale (PSS) has 18 items using a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). A composite score is calculated by adding all items (after the 7 items were reversed). A higher PSS score indicates higher stress levels.
Parental stress | One week after the intervention
  The Parental Stress Scale (PSS) has 18 items using a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). A composite score is calculated by adding all items (after the 7 items were reversed). A higher PSS score indicates higher stress levels.
Tutor efficacy for inclusive practice | One week before the intervention
  The Teacher Efficacy for Inclusive Practices scale (TEIP) is designed to measure perceived tutor efficacy in teaching in inclusive classrooms. The scale consists of 18 items scored on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). The 18 items are divided into three subscales: Efficacy to use inclusive instructions, efficacy in collaboration, and efficacy in managing behaviors.
Tutor efficacy for inclusive practice | One week after the intervention
  The Teacher Efficacy for Inclusive Practices scale (TEIP) is designed to measure perceived tutor efficacy in teaching in inclusive classrooms. The scale consists of 18 items scored on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). The 18 items are divided into three subscales: Efficacy to use inclusive instructions, efficacy in collaboration, and efficacy in managing behaviors.
Open-Ended Questions | One week before the intervention
  Open-ended questions are also included in the questionnaire to gather written feedback from the students regarding their expectations and experiences of participating in the tutoring and counseling program. Examples of open-ended questions for students include: "What difficulties have you encountered in study and life?", "What are your expectations for taking part in this tutoring and counseling program?", and "In what ways do you believe this tutoring and counseling program has been most helpful to you?". Examples of open-ended questions for tutors include: "What have you learned as a well-being tutor?", and "What are your thoughts on implementing the tutoring and counseling program for students with psychological needs?".
Open-Ended Questions | One week after the intervention
  Open-ended questions are also included in the questionnaire to gather written feedback from the students regarding their expectations and experiences of participating in the tutoring and counseling program. Examples of open-ended questions for students include: "What difficulties have you encountered in study and life?", "What are your expectations for taking part in this tutoring and counseling program?", and "In what ways do you believe this tutoring and counseling program has been most helpful to you?". Examples of open-ended questions for tutors include: "What have you learned as a well-being tutor?", and "What are your thoughts on implementing the tutoring and counseling program for students with psychological needs?".

CONTACTS AND LOCATIONS:
Locations (1):
- EdUHK, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD is not yet finalized due to ethical consideration.